CLINICAL TRIAL: NCT05585645
Title: A Multicenter, Double-blind, Randomized, Parallel Comparative Study of Efficacy and Safety of Nanogen's Darbepoetin Alfa With Aranesp® (Amgen) in the Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis
Brief Title: A Study to Compare Efficacy and Safety of Nanogen's Darbepoetin Alfa With Aranesp® (Amgen) in the Treatment of Anemia in Chronic Kidney Disease Patients on Dialysis (CKD)
Acronym: CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Collaborators: Vietstar Biomedical Research (Industry); MEDPHASE CLINICAL RESEARCH CONSULTANT COMPANY LIMITED (Unknown); CLINICAL RESEARCH VIET NAM SKILL TRAINING AND CONSULTING COMPANY LIMITED (Unknown); MedProve Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NNG06.2
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anemia; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: CKD on dialysis; Nanogen; Anemia; Darbepoetin Alfa
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimus (Experimental): NNG-DEPO (Darbepoetin alfa 10 mcg/0.4 mL, 20 mcg/0.5 mL, 40 mcg/0.4 mL, 60 mcg/0.3 mL) is available as a prefilled syringe in a sterile, colorless, glass tube.
  Storage: 2-8ºC, not frozen. The process of transporting and storing the drug must ensure the temperature in the range of 2-8ºC.
  NNG-DEPO/Aranesp is administered subcutaneously (or intravenously) at a dose of 0.75 g/kg initially, every 2 weeks at the second visit.
  Study drug will be prepared according to standard procedure (SOP). Dosage adjustment guideline:
  Patients will have hemoglobin levels monitored every 2 weeks. The investigators will evaluate and adjust the dose of Darbepoetin alfa to maintain the Hb levels within the target range (10 - 12 g/dL)
  Interventions: Biological: Stimus (NNG-DEPO)
- Aranesp (Active Comparator): Aranesp® (Darbepoetin alfa 10 mcg/ 0.4 mL, 20 mcg/ 0.5 mL, 40 mcg/ 0.4 mL, 60 mcg/ 0.3 mL) is manufactured by Amgen, as a pre-filled syringe in a sterile, glass tube, colourless.
  Storage: 2-8ºC, not frozen. The process of transporting and storing the drug must ensure the temperature in the range of 2-8ºC.
  NNG-DEPO/Aranesp is administered subcutaneously (or intravenously) at a dose of 0.75 g/kg initially, every 2 weeks at the second visit.
  Study drug will be prepared according to standard procedure (SOP). Dosage adjustment guideline:
  Patients will have hemoglobin levels monitored every 2 weeks. The investigators will evaluate and adjust the dose of Darbepoetin alfa to maintain the Hb levels within the target range (10 - 12 g/dL)
  Interventions: Biological: Stimus (NNG-DEPO)

INTERVENTIONS:
Biological: Stimus (NNG-DEPO) — Nanogen's Darbepoetin alfa 10µg/0.4mL, 20µg/0.5mL, 40µg/0.4mL, 60µg/0.3mL, prefilled syringe

SUMMARY:
This is a double-blind, two-arm, randomized, multicenter to compare the efficacy and safety of NNG-DEPO and Aranesp in CKD on dialysis patients.

Patients aged 18 to 65 years (inclusive), diagnosed with anemia due to CKD in dialysis, who meet all inclusion criteria, requiring treatment with Darbepoetin alfa. The study subjects (patients) will be randomized into a 1:1 ratio to NNG-DEPO and Aranesp treatment arms respectively. Patients will receive either NNG-DEPO or Aranesp 0.75 µg/kg by subcutaneous injection every other week for 24 weeks.

During the treatment, dose adjustments will be made as necessary to achieve a hemoglobin response, defined as maintaining Hb in the target range of 10 - 12 g/dL.

DETAILED DESCRIPTION:
The phase of the study: phase 3

Study sites:

Nguyen Tri Phuong Hospital Thu Duc City Hospital An Sinh Hospital Thong Nhat General Hospital Dong Nai

Sample size: 214 patients

TARGET POPULATION: Patients with chronic kidney disease undergoing dialysis (aged 18 to 65 years)

STUDY GROUPS:

Darbepoetin alfa (Nanogen) SC/IV route 0.75 µg/kg Q2W, for 24 weeks. Aranesp® (Amgen) SC/IV route 0.75 µg/kg Q2W, for 24 weeks.

Blood sample will be taken for Complete Blood Count (CBC) test at each visit (Week 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24) to monitor haemoglobin response.

Study Procedures:

This study was designed for 26 weeks (2 weeks for screening and 24 weeks for treatment) and there are total of 14 visits:

Visit 1 is the screening visit. Visit 2: Randomization, initiate study treatment, assess the Hb baseline. Visit 3 - 7 is to monitor, evaluate the efficacy, safety. Visit 8 is to interim assess the efficacy, safety for each patient to make the decision continous/discontinous the study treatment.

Vist 9 -13 is to monitor, evaluate the efficacy, safety. Visit 14 is termination visit.

SAFETY AND TOLERABILITY ASSESSMENT:

Safety and tolerability assessments will be performed at each visit. Following variables will be considered to define the safety and tolerability of investigational drugs:

Clinical adverse events (AEs): frequency of AEs, overall and by intensity. Severe clinical adverse events (SAEs): frequency of AEs, overall and by intensity.

Symptoms directed physical examination including body weight, and vital signs during treatment period: mean change from baseline and the frequency of clinically relevant changes from baseline.

Laboratory tests: frequency of clinically relevant changes from baseline. The frequency of any concomitant medication administered to treat any adverse events.

Presence of darbepoetin alfa anti-bodies (immunogenicity).

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the informe consent form and adhere to study visit schedule.
* Male or female patients aged from 18 to 65 years.
* Patients on hemodialysis or peritoneal dialysis for at least 3 months and have Hb baseline <10 g/dL during the screening period.
* Have transferrin saturation ≥ 20%, serum ferritin ≥ 200 ng/mL, vitamin B12 and folate within the normal range.
* Have expected survival of at least 6 months from time of enrollment (by investigator's assessment).
* Women childbearing age must agree to use medically acceptable methods of contraception during the study and for 6 months after the last study treatment.
* The patient does not have any serious medical conditions that may affect to study treatment compliance.

Exclusion Criteria:

* Uncontrolled hypertension over 2 weeks prior to and within the screening period (BP ≥ 160/90 mmHg).
* Patients treated with Darbepoetin alfa or r-HuEPO within 4 weeks prior to enrollment.
* Patients with Uncontrolled diabetes mellitus with HbA1C ≥ 10%.
* Congestive Heart Failure of grade 3 or 4 as New York Heart Association classification.
* History of unstable angina or myocardial infarction within 6 months.
* History of Grand mal seizures in last 2 years.
* Present with severe hyperparathyroidism (iPTH >1500 pg/mL for Dialysis).
* History of major surgery within 12 weeks prior to screening.
* Systemic hematologic disorders including sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma and hemolytic anemia.
* Systemic infections, active inflammatory diseases and malignancies.
* Active liver disease or hepatic with liver enzymes AST and ALT raised > 2-times of laboratory normal values, child B or child C cirrhosis.
* Are being treated with androgen therapy within the 8 weeks prior to the screening period.
* Pregnant or suspected pregnant women, breast-feeding women.
* Patients scheduled for any transplant procedure within 6 months of screening or with a previous history of kidney transplantation.
* Patients who are hypersensitive to any of substances of investigational product.
* Patients using drugs that can affect the concentration of Hb in the blood (except blood-forming drugs such as iron, folic acid).
* Patients with seropositivity to HIV, HBV or anti-HCV.
* Patients having acute tuberculosis or any acute bacterial infection within 1 month prior to the screening.
* Patient has occult blood in stool or any other known source of internal bleeding and confirmed gastrointestinal bleeding by endoscopy.
* Patients with blood transfusion due to acute bleeding within 12 weeks prior to screening period.
* Patients with a history of immunosuppressive therapy within 1 month.
* The patient is suffering from advanced cancer.
* Patients having participated in any other clinical trial within 1 month prior to the screening period.
* The patient had any medical condition that the investigator assessed as affecting the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
The mean change Hemoglobin level from baseline to Week 24 | Week 0 (Assessed predose)- Week 24

SECONDARY OUTCOMES:
Proportion of patients achieving 1 g/dL rise in Hb from baseline during 24 weeks after treatment | Week 0 (Assessed predose)- Week 24
Proportion of patients achieving Hb within the target range (10 - 12 g/dL) at week 24. | Week 24
Proportion of patients need for blood transfusion during 24 weeks after treatment. | Week 0 (Assessed predose)- Week 24
4. The mean dose of NNG-DEPO/Aranesp administered for achievement of Hb in the target Hb levels (10 - 12 g/dL) during 24 weeks. | Week 0 (Assessed predose)- Week 24
Time to initial achievement of Hb ≥ 11 g/dL. | Week 0 (Assessed predose)- Week 24
Proportion of the adverse events (AE) including physical examinations, vital signs, and clinical laboratory investigations. | Week 0 (Assessed predose)- Week 24
Proportion of patients positive with anti-Darbepoetin alfa antibody after treatment. | Week 0 (Assessed predose)- Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bui V Pham, MD. PhD, Principal Investigator — Nguyen Tri Phuong Hospital
Locations (1):
- NANOGEN Pharmaceutical Biotechnology JSC, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
Not yet infomation